CLINICAL TRIAL: NCT06134297
Title: Adherence, Feasibility, Clinical Evolution Therapeutic Efficacy of Three Different Muscle Overload Models Used for Physical Rehabilitation of Patients Undergoing Bone Marrow Transplantation: a Randomized Clinical Trial
Brief Title: Adherence, Viability, Clinical Evolution and Therapeutic Efficacy in Patients Undergoing Bone Marrow Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 54240221.5.0000.5335
Record Dates: First submitted 2023-10-16; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stem Cell Transplantation
Keywords: Exercise Therapy; Fatigue; Hematologic Neoplasms
MeSH Terms: conditions — Fatigue; Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Group (Experimental): Aerobic exercise using a cycle ergometer lasting 15 consecutive minutes with load adjusted to maintain heart rate (HR) between 65-75% of the maximum HR predicted for age (HRmax = 200-age).
  Interventions: Device: Cycle ergometer
- Anaerobic Exercise Group (Experimental): Muscle strength training using shin guards and elastic bands to promote muscle overload, generating maximum force production, where the contraction time should not exceed 20 seconds.
  Interventions: Device: Strength Training - elastic band and shin guards
- Mixed Exercise Group (Experimental): Exercises through alternation between aerobic and anaerobic overload (performing the exercises from the previously mentioned groups on alternate days), in a 1:1 ratio until the end of the physical rehabilitation program.
  Interventions: Device: Cycle ergometer, elastic band and shin guards

INTERVENTIONS:
Device: Cycle ergometer — The Aerobic Exercise Group will perform a cycle ergometer for 15 consecutive minutes with a load adjusted to maintain heart rate (HR) between 65-75% of the maximum HR predicted for age (HRmax = 200-age). Peripheral oxygen saturation will be controlled and, upon a sustained drop (> 2 minutes after load reduction) below 90%, the session will be interrupted. The subjective feeling of tiredness in the legs and shortness of breath will be constantly monitored and if values equal to or greater than 8 (0-10) occur, the exercise will be stopped.
  Arms: Aerobic Exercise Group
Device: Strength Training - elastic band and shin guards — The Anaerobic Exercise Group will perform muscular strength training using maximum strength, where the contraction time should not exceed 20 seconds. For the upper limbs, the overload used will be through the use of an elastic band, with guidance for the patient to perform the shoulder external rotation exercise, elbow flexion exercises and open row rowing exercise. For the lower limbs, bridge movements, lunges and sit-up exercises will be performed with a maximum of 15 repetitions, and overload with ankle weights or dumbbells can be used in addition to body weight. The muscle contraction should lead the patient to a state of muscular fatigue and if the objective is not achieved, the exercise will be adapted to require greater strength from the patient so that he or she can reach maximum strength.
  Arms: Anaerobic Exercise Group
Device: Cycle ergometer, elastic band and shin guards — Mixed Exercise Group will perform the exercises by alternating between aerobic and anaerobic overload, in a 1:1 ratio until the end of the physical rehabilitation program, following exactly the same protocols described previously (alternating one session of the aerobic protocol and in the following session the anaerobic protocol).
  Arms: Mixed Exercise Group

SUMMARY:
Hematological neoplasms originate from the differentiation and proliferation of abnormal lymphatic or myeloid cells that alter the constitution of elements of the blood, bone marrow and lymph nodes. Treatment includes high-dose chemotherapy alone or associated with hematopoietic stem cell transplantation (HSCT). However, the adverse effects of this treatment affect multiple organs and systems, reducing physical capacity, increasing the feeling of fatigue, anxiety and depression, which together affect quality of life. Patients who exercise before, during or after anti-neoplastic treatment demonstrate significant benefits. But rehabilitating physical capacity involves the challenge of fluctuations in the patient's readiness along with daily clinical variations, which ultimately directly affects the rate of adherence to exercises, impacting the effectiveness of the physical rehabilitation program. There is no specific individualization of muscular overload that takes into account such variability in pathophysiological, functional and psychological situations, but the cardiorespiratory response and muscular strength performance in the face of progressive overload can be measured with sufficient recovery periods to optimize the physiological adaptations promoted by muscular overload. regularly, even in patients undergoing antineoplastic treatment. Objective: To evaluate the adherence rate, operational feasibility, clinical/behavioral evolution and effectiveness of three different muscle overload models (aerobic, anaerobic and mixed) used for the physical rehabilitation of patients hospitalized for antineoplastic hematological treatment with HSCT

DETAILED DESCRIPTION:
This is a randomized clinical trial. Patients will be allocated into groups (1) Aerobic; (2) Anaerobic and (3) Mixed. The manifestation of signs and symptoms will be evaluated using the Edmonton Symptom Assessment System (ESAS) inventory, a sensation of fatigue using the multidimensional fatigue questionnaire (MIF), and quality of life using the European Organization for Research and Treatment of Cancer Core Quality of Life questionnaire. Questionnaire (EORTC QLQ-30) and the incidence and intensity of anxiety and depression symptoms using the General Hospital Anxiety and Depression Scale (HAD), in addition to the strength assessment of the upper limbs (HANDGRIP) and lower limbs (TSL). Participants in the aerobic group will perform exercises for the lower limbs with a cycle ergometer for 15 consecutive minutes and participants in the anaerobic group will perform exercises with an overload of shin weights or dumbbells of 0.5kg/1kg for large muscle groups. Participants in the mixed group will have a mixed muscular overload, performed by alternating between aerobic and anaerobic overload with a 1:1 ratio until the end of the program.

ELIGIBILITY:
Inclusion criteria:

* Be between 18 and 64 years old;
* Present hematological malignancy undergoing first antineoplastic treatment with HSCT;
* Have intact neurological function and cognition;
* Be in clinical conditions that allow participation in physical rehabilitation;
* To agree with the study proposal by signing the Free and Informed Consent Form (TCLE).

Exclusion criteria:

* Present clinical complications that impair the performance of motor physiotherapy, including the practice of cycle ergometer and resistance exercises;
* Present previous musculoskeletal changes that interfere with the execution of physical performance assessment tests;
* Patients with limiting cardiovascular or pulmonary disease, significant psychiatric or neurological disorders and/or limiting interpretation of documents and forms that will be used in the study;
* Patients who require mobility assistance and/or diagnosed with multiple myeloma with or without the presence of bone metastasis;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the physical rehabilitation program for lower limb strength through sitting and standing exercises | During the period of hospital stay, an average 1 month.
  It will be determined by evaluating lower limb strength performance in the 30-second sit-to-stand test. The score will be based on the number of repetitions performed during the 30 timed seconds.
Effectiveness of the physical rehabilitation program for upper limb strength using dynamometry | During the period of hospital stay, an average 1 month
  It will be determined by evaluating the strength performance of the upper limbs through dynamometry. The value will be given in kilograms of force. And it will be calculated through the average of three measurements.
Adherence to physical rehabilitation sessions | During the period of hospital stay, an average 1 month
  It will be evaluated through the ratio between the number of sessions actually carried out by the number of days in which the minimum clinical conditions for practicing physical exercise can be fully characterized during the hospital admission.
Operational viability for implementing the exercise protocol | During the period of hospital stay, an average 1 month
  It will be evaluated through the time needed to execute the different muscle overload protocols
Satisfaction with physiotherapy care | During the period of hospital stay, an average 1 month
  It will be evaluated through a satisfaction questionnaire (contains 11 questions and a maximum score of 55 points; the higher the score, the better the test result and better satisfaction).
Clinical behavioral evolution of signs and symptoms related to cancer | During the period of hospital stay, an average 1 month
  The following will be carried out at the beginning and end of the intervention:
  - Edmonton Sympton Assessment System Inventory (scale with 9 items; each can be scored from 0 to 10; the final value of the scale is the sum of each item; the higher the score, the worse the symptoms).
Clinical behavioral evolution of signs of fatigue | During the period of hospital stay, an average 1 month
  The following will be carried out at the beginning and end of the intervention:
  - Multidimensional Fatigue Questionnaire - (20 questions scored from 1 to 5; the higher the final score, the worse the symptoms).
Clinical behavioral evolution of signs of anxiety and depression | During the period of hospital stay, an average 1 month
  The following will be carried out at the beginning and end of the intervention:
  - General Hospital Anxiety and Depression Scale (14 questions, scored from 0 to 3; the higher the final score, the worse the symptoms).
Clinical behavioral evolution of quality of life perception | During the period of hospital stay, an average 1 month
  The following will be carried out at the beginning and end of the intervention:
  - Basic Quality of Life Questionnaire of the European Organization for Research and Treatment of Cancer (30 questions scored from 1 to 4; the higher the final score, the worse the symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio E Macagnan, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wehrle A, Kneis S, Dickhuth HH, Gollhofer A, Bertz H. Endurance and resistance training in patients with acute leukemia undergoing induction chemotherapy-a randomized pilot study. Support Care Cancer. 2019 Mar;27(3):1071-1079. doi: 10.1007/s00520-018-4396-6. Epub 2018 Aug 18. PMID 30121789
- [Background] van Haren IE, Timmerman H, Potting CM, Blijlevens NM, Staal JB, Nijhuis-van der Sanden MW. Physical exercise for patients undergoing hematopoietic stem cell transplantation: systematic review and meta-analyses of randomized controlled trials. Phys Ther. 2013 Apr;93(4):514-28. doi: 10.2522/ptj.20120181. Epub 2012 Dec 6. PMID 23224217
- [Background] Tran J, Norder EE, Diaz PT, Phillips GS, Elder P, Devine SM, Wood KL. Pulmonary rehabilitation for bronchiolitis obliterans syndrome after hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2012 Aug;18(8):1250-4. doi: 10.1016/j.bbmt.2012.01.017. Epub 2012 Jan 30. PMID 22300617
- [Background] THOMAS ED, LOCHTE HL Jr, CANNON JH, SAHLER OD, FERREBEE JW. Supralethal whole body irradiation and isologous marrow transplantation in man. J Clin Invest. 1959 Oct;38(10 Pt 1-2):1709-16. doi: 10.1172/JCI103949. No abstract available. PMID 13837954
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Steinberg A, Asher A, Bailey C, Fu JB. The role of physical rehabilitation in stem cell transplantation patients. Support Care Cancer. 2015 Aug;23(8):2447-60. doi: 10.1007/s00520-015-2744-3. Epub 2015 May 14. PMID 25971213
- [Background] Storb R, Sandmaier BM. Nonmyeloablative allogeneic hematopoietic cell transplantation. Haematologica. 2016 May;101(5):521-30. doi: 10.3324/haematol.2015.132860. PMID 27132278
- [Background] de Souza CV, Miranda EC, Garcia C Jr, Aranha FJ, de Souza CA, Vigorito AC. Functional evaluation indicates physical losses after hematopoietic stem cell transplantation. Rev Bras Hematol Hemoter. 2012;34(5):345-51. doi: 10.5581/1516-8484.20120090. PMID 23125542
- [Background] Shechtman O, Sindhu BS, Davenport PW. Using the force-time curve to detect maximal grip strength effort. J Hand Ther. 2007 Jan-Mar;20(1):37-47; quiz 48. doi: 10.1197/j.jht.2006.10.006. PMID 17254907
- [Background] Schuler MK, Hornemann B, Pawandenat C, Kramer M, Hentschel L, Beck H, Kasten P, Singer S, Schaich M, Ehninger G, Platzbecker U, Schetelig J, Bornhauser M. Feasibility of an exercise programme in elderly patients undergoing allogeneic stem cell transplantation - a pilot study. Eur J Cancer Care (Engl). 2016 Sep;25(5):839-48. doi: 10.1111/ecc.12400. Epub 2015 Nov 3. PMID 26526286
- [Background] Sasso JP, Eves ND, Christensen JF, Koelwyn GJ, Scott J, Jones LW. A framework for prescription in exercise-oncology research. J Cachexia Sarcopenia Muscle. 2015 Jun;6(2):115-24. doi: 10.1002/jcsm.12042. Epub 2015 May 11. PMID 26136187
- [Background] Ries AL, Make BJ, Lee SM, Krasna MJ, Bartels M, Crouch R, Fishman AP; National Emphysema Treatment Trial Research Group. The effects of pulmonary rehabilitation in the national emphysema treatment trial. Chest. 2005 Dec;128(6):3799-809. doi: 10.1378/chest.128.6.3799. PMID 16354848
- [Background] van Dongen JM, Persoon S, Jongeneel G, Bosmans JE, Kersten MJ, Brug J, Nollet F, Chinapaw MJM, Buffart LM. Long-term effectiveness and cost-effectiveness of an 18-week supervised exercise program in patients treated with autologous stem cell transplantation: results from the EXIST study. J Cancer Surviv. 2019 Aug;13(4):558-569. doi: 10.1007/s11764-019-00775-9. Epub 2019 Jul 8. PMID 31286387
- [Background] Persoon S, Kersten MJ, van der Weiden K, Buffart LM, Nollet F, Brug J, Chinapaw MJ. Effects of exercise in patients treated with stem cell transplantation for a hematologic malignancy: a systematic review and meta-analysis. Cancer Treat Rev. 2013 Oct;39(6):682-90. doi: 10.1016/j.ctrv.2013.01.001. Epub 2013 Feb 26. PMID 23485478
- [Background] Paul KL. Rehabilitation and exercise considerations in hematologic malignancies. Am J Phys Med Rehabil. 2011 May;90(5 Suppl 1):S88-94. doi: 10.1097/PHM.0b013e31820be055. PMID 21765268
- [Background] Oechsle K, Aslan Z, Suesse Y, Jensen W, Bokemeyer C, de Wit M. Multimodal exercise training during myeloablative chemotherapy: a prospective randomized pilot trial. Support Care Cancer. 2014 Jan;22(1):63-9. doi: 10.1007/s00520-013-1927-z. Epub 2013 Aug 29. PMID 23989498
- [Background] Mosher CE, Redd WH, Rini CM, Burkhalter JE, DuHamel KN. Physical, psychological, and social sequelae following hematopoietic stem cell transplantation: a review of the literature. Psychooncology. 2009 Feb;18(2):113-27. doi: 10.1002/pon.1399. PMID 18677717
- [Background] Morishita S, Kaida K, Yamauchi S, Wakasugi T, Ikegame K, Ogawa H, Domen K. Relationship of physical activity with physical function and health-related quality of life in patients having undergone allogeneic haematopoietic stem-cell transplantation. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12669. Epub 2017 Feb 21. PMID 28220548
- [Background] Morishita S, Kaida K, Setogawa K, Kajihara K, Ishii S, Ikegame K, Kodama N, Ogawa H, Domen K. Safety and feasibility of physical therapy in cytopenic patients during allogeneic haematopoietic stem cell transplantation. Eur J Cancer Care (Engl). 2013 May;22(3):289-99. doi: 10.1111/ecc.12027. Epub 2012 Dec 18. PMID 23252444
- [Background] Mancuso EV, Rezende NA. [Pulmonary function testing in bone marrow transplantation: a systematic review]. Rev Port Pneumol. 2006 Jan-Feb;12(1):61-9. doi: 10.1016/s0873-2159(15)30422-0. Portuguese. PMID 16572257
- [Background] Liu RD, Chinapaw MJ, Huijgens PC, van Mechelen W. Physical exercise interventions in haematological cancer patients, feasible to conduct but effectiveness to be established: a systematic literature review. Cancer Treat Rev. 2009 Apr;35(2):185-92. doi: 10.1016/j.ctrv.2008.09.008. Epub 2008 Nov 11. PMID 19004560
- [Background] Kuehl R, Schmidt ME, Dreger P, Steindorf K, Bohus M, Wiskemann J. Determinants of exercise adherence and contamination in a randomized controlled trial in cancer patients during and after allogeneic HCT. Support Care Cancer. 2016 Oct;24(10):4327-37. doi: 10.1007/s00520-016-3271-6. Epub 2016 May 17. PMID 27189616
- [Background] Knips L, Bergenthal N, Streckmann F, Monsef I, Elter T, Skoetz N. Aerobic physical exercise for adult patients with haematological malignancies. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD009075. doi: 10.1002/14651858.CD009075.pub3. PMID 30702150
- [Background] Kovalszki A, Schumaker GL, Klein A, Terrin N, White AC. Reduced respiratory and skeletal muscle strength in survivors of sibling or unrelated donor hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Jun;41(11):965-9. doi: 10.1038/bmt.2008.15. Epub 2008 Feb 11. PMID 18264142
- [Background] Kawada S, Kobayashi K, Ohtani M, Fukusaki C. Cystine and theanine supplementation restores high-intensity resistance exercise-induced attenuation of natural killer cell activity in well-trained men. J Strength Cond Res. 2010 Mar;24(3):846-51. doi: 10.1519/JSC.0b013e3181c7c299. PMID 20145562
- [Background] Jarden M, Baadsgaard MT, Hovgaard DJ, Boesen E, Adamsen L. A randomized trial on the effect of a multimodal intervention on physical capacity, functional performance and quality of life in adult patients undergoing allogeneic SCT. Bone Marrow Transplant. 2009 May;43(9):725-37. doi: 10.1038/bmt.2009.27. Epub 2009 Feb 23. PMID 19234513
- [Background] Hacker ED, Larson J, Kujath A, Peace D, Rondelli D, Gaston L. Strength training following hematopoietic stem cell transplantation. Cancer Nurs. 2011 May-Jun;34(3):238-49. doi: 10.1097/NCC.0b013e3181fb3686. PMID 21116175
- [Background] Gratwohl A, Baldomero H, Horisberger B, Schmid C, Passweg J, Urbano-Ispizua A; Accreditation Committee of the European Group for Blood and Marrow Transplantation (EBMT). Current trends in hematopoietic stem cell transplantation in Europe. Blood. 2002 Oct 1;100(7):2374-86. doi: 10.1182/blood-2002-03-0675. PMID 12239145
- [Background] Fairman CM, Zourdos MC, Helms ER, Focht BC. A Scientific Rationale to Improve Resistance Training Prescription in Exercise Oncology. Sports Med. 2017 Aug;47(8):1457-1465. doi: 10.1007/s40279-017-0673-7. PMID 28074412
- [Background] Elter T, Stipanov M, Heuser E, von Bergwelt-Baildon M, Bloch W, Hallek M, Baumann F. Is physical exercise possible in patients with critical cytopenia undergoing intensive chemotherapy for acute leukaemia or aggressive lymphoma? Int J Hematol. 2009 Sep;90(2):199-204. doi: 10.1007/s12185-009-0376-4. Epub 2009 Jul 24. PMID 19629631
- [Background] Duregon F, Gobbo S, Bullo V, Roma E, Vendramin B, Bergamo M, Bocalini DS, Di Blasio A, Cugusi L, Neunhaeuserer D, Bergamin M, Ermolao A. Exercise prescription and tailored physical activity intervention in onco-hematology inpatients, a personalized bedside approach to improve clinical best practice. Hematol Oncol. 2019 Aug;37(3):277-284. doi: 10.1002/hon.2576. Epub 2019 Mar 18. PMID 30736102
- [Background] Dimeo F, Schwartz S, Fietz T, Wanjura T, Boning D, Thiel E. Effects of endurance training on the physical performance of patients with hematological malignancies during chemotherapy. Support Care Cancer. 2003 Oct;11(10):623-8. doi: 10.1007/s00520-003-0512-2. Epub 2003 Aug 26. PMID 12942360
- [Background] Cunningham BA, Morris G, Cheney CL, Buergel N, Aker SN, Lenssen P. Effects of resistive exercise on skeletal muscle in marrow transplant recipients receiving total parenteral nutrition. JPEN J Parenter Enteral Nutr. 1986 Nov-Dec;10(6):558-63. doi: 10.1177/0148607186010006558. PMID 3098997
- [Background] Cullen M. 'Best supportive care' has had its day. Lancet Oncol. 2001 Mar;2(3):173-5. doi: 10.1016/S1470-2045(00)00260-6. PMID 11902569
- [Background] Courneya KS, Keats MR, Turner AR. Physical exercise and quality of life in cancer patients following high dose chemotherapy and autologous bone marrow transplantation. Psychooncology. 2000 Mar-Apr;9(2):127-36. doi: 10.1002/(sici)1099-1611(200003/04)9:23.0.co;2-l. PMID 10767750
- [Background] Chang PH, Lai YH, Shun SC, Lin LY, Chen ML, Yang Y, Tsai JC, Huang GS, Cheng SY. Effects of a walking intervention on fatigue-related experiences of hospitalized acute myelogenous leukemia patients undergoing chemotherapy: a randomized controlled trial. J Pain Symptom Manage. 2008 May;35(5):524-34. doi: 10.1016/j.jpainsymman.2007.06.013. Epub 2008 Feb 15. PMID 18280104
- [Background] Castro MM, Quarantini L, Batista-Neves S, Kraychete DC, Daltro C, Miranda-Scippa A. [Validity of the hospital anxiety and depression scale in patients with chronic pain.]. Rev Bras Anestesiol. 2006 Oct;56(5):470-7. doi: 10.1590/s0034-70942006000500005. Portuguese. PMID 19468593
- [Background] Carlson LE, Smith D, Russell J, Fibich C, Whittaker T. Individualized exercise program for the treatment of severe fatigue in patients after allogeneic hematopoietic stem-cell transplant: a pilot study. Bone Marrow Transplant. 2006 May;37(10):945-54. doi: 10.1038/sj.bmt.1705343. PMID 16565742
- [Background] Bewarder M, Klostermann A, Ahlgrimm M, Bittenbring JT, Pfreundschuh M, Wagenpfeil S, Kaddu-Mulindwa D. Safety and feasibility of electrical muscle stimulation in patients undergoing autologous and allogeneic stem cell transplantation or intensive chemotherapy. Support Care Cancer. 2019 Mar;27(3):1013-1020. doi: 10.1007/s00520-018-4390-z. Epub 2018 Aug 9. PMID 30094730
- [Background] Bergenthal N, Will A, Streckmann F, Wolkewitz KD, Monsef I, Engert A, Elter T, Skoetz N. Aerobic physical exercise for adult patients with haematological malignancies. Cochrane Database Syst Rev. 2014 Nov 11;(11):CD009075. doi: 10.1002/14651858.CD009075.pub2. PMID 25386666
- [Background] Baumann FT, Zopf EM, Nykamp E, Kraut L, Schule K, Elter T, Fauser AA, Bloch W. Physical activity for patients undergoing an allogeneic hematopoietic stem cell transplantation: benefits of a moderate exercise intervention. Eur J Haematol. 2011 Aug;87(2):148-56. doi: 10.1111/j.1600-0609.2011.01640.x. PMID 21545527
- [Background] Afessa B, Peters SG. Chronic lung disease after hematopoietic stem cell transplantation. Clin Chest Med. 2005 Dec;26(4):571-86, vi. doi: 10.1016/j.ccm.2005.06.012. PMID 16263397